CLINICAL TRIAL: NCT01739140
Title: Yoga for Chronic Low Back Pain and Its Mechanism of Action (YoMA)
Acronym: YoMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Bowes Fund for Innovative Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSFCHR12-09424
Record Dates: First submitted 2012-11-27; First posted 2012-12-03 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Yoga (Experimental): Study Participants will receive: 12 weekly yoga classes, a book and a home practice audio recording.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga

SUMMARY:
This is a study to better understand how a yoga intervention helps improve symptoms in people with chronic low back pain. This study will be a 12-week intervention of about 24 participants with chronic low back pain where all individuals will receive weekly yoga classes and instructions for home practice. The purpose of this study is to collect feasibility data and to conduct preliminary analyses in preparation for a larger planned NIH study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain lasting > 3 months
* Back pain that is rated at least 3 on a numeric pain rating scale that ranges from 0 to 10 (0-no pain, 10 worst pain imaginable).
* English language fluency

Exclusion Criteria:

* BMI > 40
* Inability to provide informed consent
* Recent diagnosis of abdominal aneurism
* Recent diagnosis of metastatic cancer
* Recent diagnosis of discitis
* Recent diagnosis of disk disease
* Recent diagnosis of spinal stenosis
* Recent diagnosis of spondylolisthesis
* Recent diagnosis of infectious cause of back pain
* Recent diagnosis of fracture of vertebra
* Recent diagnosis of Fibromyalgia
* Recent diagnosis of rheumatoid arthritis
* Recent diagnosis of ankylosing spondylitis
* Recent diagnosis of paralysis
* Pregnancy
* Prior or planned back surgery
* Blindness or severe vision problems
* Deafness or severe hearing problems
* Bipolar or manic depression and not taking medication
* Major depression
* Psychoses (major)
* a substance abuse condition
* Dementia
* Unable to get up and down from the floor
* Involvement in a lawsuit related to back pain
* Lack of transportation
* Other disabling chronic conditions (e.g., disabling heart or lung disease, diabetic neuropathy, receiving treatment for hepatitis)
* Currently (within the past 3 months) using yoga classes for more than 15 minutes per week
* Inability to be contacted by phone or email
* no computer access
* schedule does not allow for participation in classes/home practice
* planning to move out of town or take a long vacation during the period of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire | Baseline to 3 months post-intervention.

SECONDARY OUTCOMES:
Numeric Rating Scale for Pain | Baseline to 3 months post-intervention.
Pain Medication Usage Survey | Baseline to 3 months post-intervention.

OTHER OUTCOMES:
Inflammatory pain related cytokines | Baseline to 3 months post-intervention.
Heart rate variability | Baseline to 3 months post-intervention.
International Physical Activity Questionnaire | Baseline to 3 months post-intervention.
Pain Catastrophizing Scale | Baseline to 3 months post-intervention.
Five Facet Mindfulness Questionnaire | Baseline to 3 months post-intervention.
Multidimensional Assessment of Interoceptive Awareness | Baseline to 3 months post-intervention.
Patient Reported Outcomes Measurement Information System: Pain - Behavior | Baseline to 3 months post-intervention.
Patient Reported Outcomes Measurement Information System: Pain - Interference | Baseline to 3 months post-intervention.
Patient Reported Outcomes Measurement Information System: Emotional Distress - Depression | Baseline to 3 months post-intervention.
Patient Reported Outcomes Measurement Information System: Emotional Distress - Anxiety | Baseline to 3 months post-intervention.
Patient Reported Outcomes Measurement Information System: Physical Function | Baseline to 3 months post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Corey, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco's Osher Center for Integrative Medicine, San Francisco, California, United States